CLINICAL TRIAL: NCT00432458
Title: A Phase III Randomized Trial of Thalidomide Plus Zoledronic Acid Versus Zoledronic Acid Alone in Patients With Early Stage Multiple Myeloma
Brief Title: Zoledronate With or Without Thalidomide in Treating Patients With Early Stage Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000530050; P30CA015083 (NIH); MC0289 (Other: Mayo Clinic Cancer Center); 421-03 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2007-02-05; First posted 2007-02-07 (Estimated); Results first posted 2012-07-04 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-06

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Thalidomide; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: Thal/ZLD (Experimental): Thalidomide (Thal) + Zolendronic acid (ZLD)
  Interventions: Drug: Thalidomide; Drug: zoledronic acid
- Arm II: ZLD (Experimental): Zoledronic acid (ZLD)
  Interventions: Drug: zoledronic acid

INTERVENTIONS:
Drug: Thalidomide — 200 mg orally on days 1-28 of 28 day cycle
  Arms: Arm I: Thal/ZLD
Drug: zoledronic acid — 4 mg^2 by IV on day 1 every 84 days for 1 year and once per year thereafter

SUMMARY:
RATIONALE: Zoledronate may prevent bone loss and stop the growth of cancer cells in bone. Thalidomide may stop the growth of cancer cells by blocking blood flow to the cancer. It is not yet know whether giving zoledronate together with thalidomide is more effective than zoledronate alone in treating multiple myeloma.

PURPOSE: This randomized phase III trial is studying zoledronate and thalidomide see how well they work compared with zoledronate alone in treating patients with early stage multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare time to progression in patients with early stage multiple myeloma treated with zoledronate with or without thalidomide.

Secondary

* Compare the response rate, 1-year progression-free survival rate, duration of response, and time to next therapy in patients treated with these regimens.
* Assess differences in toxicity of these regimens in these patients.

OUTLINE: This is a multicenter, randomized study. Patients are stratified according to the presence of lytic lesions on metastatic bone survey (yes vs no), beta-2 microglobulin level (high vs normal), and bone marrow labeling index (high [> 1.0%] vs low [≤ 1.0%]). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral thalidomide on days 1-28. Treatment with thalidomide repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive zoledronate IV over 15 minutes on day 1. Treatment with zoledronate repeats every 84 days for 1 year and once a year thereafter in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive zoledronate IV over 15 minutes on day 1. Treatment repeats every 84 days for 1 year and once a year thereafter in the absence of disease progression or unacceptable toxicity.

Blood samples are collected for research studies at baseline and after courses 3, 6, 9, and 12. Bone marrow aspirates are performed at baseline and after courses 6 and 12. Samples are evaluated for bone marrow angiogenesis; vascular endothelial growth factor (VEGF), VEGF receptor 1 (VEGFR-1), and VEGFR-2 expression; bone marrow angiogenesis-VEGF relationship; bone marrow angiogenesis/apoptosis rate relationship; bone marrow angiogenesis/plasma cell (PC) proliferation rate relationship; VEGF expression/apoptosis rate relationship; and VEGFR expression/PC proliferation rate relationship.

After completion of study treatment, patients are followed every 6 months for up to 5 years.

PROJECTED ACCRUAL: A total of 120 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma (MM)

  * Previously untreated asymptomatic disease
  * No requirement for immediate chemotherapy for active MM, such as hypercalcemia from myeloma or painful bone lesions
* No solitary plasmacytoma
* Measurable or evaluable disease as defined by one of the following:

  * Serum monoclonal protein ≥ 1.0 g by protein electrophoresis
  * More than 200 mg of monoclonal protein in the urine by 24-hour electrophoresis
  * Measurable soft tissue plasmacytoma by physical exam with ruler or by MRI or positron emission tomography/CT scan

    * If the only measurable lesion is the plasmacytoma, it must be ≥ 1.5 cm in 1 dimension
* Must have ≥ 10% plasma cells as measured on the bone marrow aspirate, bone marrow biopsy, or labeling index
* No amyloidosis

PATIENT CHARACTERISTICS:

* Performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 8.0 g/dL
* Creatinine ≤ 2.0 mg/dL (elevation above normal range should not be felt to be related to myeloma)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 methods of effective contraception 4 weeks before, during, and for 4 weeks after completion of study treatment
* No uncontrolled infection
* No other active malignancy
* No New York Heart Association class III or IV heart disease
* No pre-existing neuropathy ≥ grade 2
* No concurrent major dental work

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior corticosteroids (for nonmalignant disorders) allowed
* Prior therapy with experimental agents not shown to have significant activity in MM, such as clarithromycin, dehydroepiandrosterone, and anakinra allowed
* No prior thalidomide or corticosteroids for MM
* No more than 3 doses of IV zoledronate or pamidronate within the past 12 months
* At least 3 months since prior radiotherapy, including radiotherapy for solitary plasmacytoma
* No concurrent oral bisphosphonate therapy for osteoporosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2003-07; Primary Completion 2011-06 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Witzig, MD, Study Chair — Mayo Clinic; Craig Reeder, M.D., Principal Investigator — Mayo Clinic; Vivek Roy, M.D., Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Witzig TE, Laumann KM, Lacy MQ, Hayman SR, Dispenzieri A, Kumar S, Reeder CB, Roy V, Lust JA, Gertz MA, Greipp PR, Hassoun H, Mandrekar SJ, Rajkumar SV. A phase III randomized trial of thalidomide plus zoledronic acid versus zoledronic acid alone in patients with asymptomatic multiple myeloma. Leukemia. 2013 Jan;27(1):220-5. doi: 10.1038/leu.2012.236. Epub 2012 Aug 20. PMID 22902362

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty-eight (68) participants were recruited at Mayo Clinic (Rochester) and Memorial Sloan-Kettering between July 2003 and March 2009.
Pre-assignment Details: All 68 participants were randomized.
Period: Overall Study
Arm/Group | Arm I: Thal/ZLD | Arm II: ZLD
Started | 35 | 33
Completed | 30 | 32
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Thal/ZLD | Arm II: ZLD | Total
Number analyzed (Participants) | 35 | 33 | 68
Age Continuous [Median (Full Range); unit: years] | 63 [47 to 84] | 63 [47 to 80] | 63 [47 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 22 | 19 | 41
Region of Enrollment [Number; unit: participants]
  United States | 35 | 33 | 68
Beta-2 Microglobulin [Number; unit: participants] — The upper limit of normal for Beta-2 microglobulin was 1.80 mcg/mL.
  participants
    High (> upper limit of normal) | 29 | 26 | 55
    Normal (<= upper limit of normal) | 6 | 7 | 13
Lytic Bone Lesions [Number; unit: participants]
  Present | 2 | 2 | 4
  Not Present | 33 | 31 | 64
Bone Marrow Labeling Index [Number; unit: participants] — The labeling index indicates how fast the cancer cells are growing. This test is done in specialized labs, using myeloma cells from bone marrow samples. A high labeling index can predict a more rapid accumulation of cancer cells and a worse outlook.
  participants
    High (> 1.0%) | 3 | 3 | 6
    Low (<= 1.0%) | 31 | 30 | 61
    Not Applicable | 1 | 0 | 1
Anemia [Number; unit: participants] — The lower limit of normal (LLN) is institution specific, typically about 13.5 g/dL for males and 12.0 g/dL for females.
  participants
    < lower limit of normal | 14 | 18 | 32
    >= lower limit of normal | 21 | 15 | 36
Peripheral blood circulating plasma cells [Number; unit: participants] — Peripheral blood circulating plasma cells are cells which live outside of the bone marrow.
  participants
    Yes | 13 | 14 | 27
    No | 20 | 18 | 38
    Not Applicable | 1 | 0 | 1
    Not Done | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Progression (TTP)
Description: Time to disease progression (TTP) was defined as the time from randomization to the earliest documentation of disease progression. Participants were followed for a maximum of 5 years from registration. The median OS with 95% CI was estimated using the Kaplan Meier method, a two-sided (stratified) log-rank test was calculated.
Time Frame: randomization to progression (up to 5 years)
Population: Time to disease progression was analyzed on all randomized participants on an intent to treat basis.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm I: Thal/ZLD | Arm II: ZLD
Number analyzed (Participants) | 35 | 33
years | 2.4 [1.4 to 3.6] | 1.2 [0.7 to 2.5]
Statistical Analysis 1: Comparison: Arm I: Thal/ZLD vs Arm II: ZLD; Test type: Superiority or Other; p = 0.02, Log Rank; Model was stratified by beta-2 microglobulin (high vs low), lytic bone lesions (present vs not) and bone marrow labeling index (high vs low)

2. Secondary Outcome: 12-month Progression-free Survival (PFS)
Description: PFS at 12 months is a dichotomized outcome indicating whether or not a participant was progression free (and alive) at 12 months from the date of randomization.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Arm I: Thal/ZLD | Arm II: ZLD
Number analyzed (Participants) | 35 | 33
participants | 30 | 18
Statistical Analysis 1: Comparison: Arm I: Thal/ZLD vs Arm II: ZLD; Test type: Superiority or Other; p = 0.0048, Chi-squared

3. Secondary Outcome: Number of Participants With a Confirmed Response (Complete Response [CR], Very Good Partial Response [VGPR] or Partial Response [PR]) on Two Consecutive Evaluations at Least 2 Weeks Apart in the First 12 Months of Treatment
Description: Response is defined as follows:
  * CR: Complete disappearance of M-protein from serum & urine on immunofixation, <5% plasma cells in bone marrow (BM)
  * VGPR: >=90% reduction in serum M-component; Urine M-Component <100 mg per 24 hours; <=5% plasma cells in BM
  * PR: >= 50% reduction in serum M-Component and/or Urine M-Component >= 90% reduction or <200 mg per 24 hours; or >= 50% decrease in difference between involved and uninvolved FLC levels
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Arm I: Thal/ZLD | Arm II: ZLD
Number analyzed (Participants) | 35 | 33
participants | 13 | 0
Statistical Analysis 1: Comparison: Arm I: Thal/ZLD vs Arm II: ZLD; Test type: Superiority or Other; p < 0.001, Chi-squared

4. Secondary Outcome: Duration of Response (Complete Response, Partial Response, and Very Good Partial Response)
Description: Duration of response (DOR) is defined as the time from first documentation of response (CR, VGPR or PR) to disease progression. The median DOR with 95% CI was estimated using the Kaplan Meier method
Time Frame: time from start of response to progression (up to 5 years)
Population: Participants who achieved a confirmed response (CR, VGPR, or PR) as described above were analyzed.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm I: Thal/ZLD | Arm II: ZLD
Number analyzed (Participants) | 13 | 0
years | 3.3 [1.1 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event at the final time point for assessment |

5. Secondary Outcome: Time to Subsequent Treatment
Description: Time to subsequent treatment (TTS) was defined as time from end of active (protocol) treatment to the start of subsequent treatment for participants with progressive disease. The median TTS with 95% CI was estimated using the Kaplan Meier method
Time Frame: time from end of treatment to subsequent treatment (up to 5 years)
Population: This data was not (and will never be) analyzed as it was not submitted consistently across all participants.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm I: Thal/ZLD | Arm II: ZLD
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure (TTF) was defined as the time from randomization to the date at which the patient was removed from (protocol) treatment due to disease progression, unacceptable toxicity, participant refusal or death. The median TTF with 95% CI was estimated using the Kaplan Meier method
Time Frame: time from randomization to treatment failure (up to 5 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I: Thal/ZLD | Arm II: ZLD
Number analyzed (Participants) | 35 | 33
months | 16.5 [9.5 to 27.6] | 11.1 [8.4 to 16.7]

7. Secondary Outcome: Number of Participants With Severe (Grade 3, 4 or 5) Adverse Events
Description: Adverse events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 2.
  Description of Grades:
  Grade 1: Mild Grade 2: Moderate Grade 3: Severe Grade 4: Life-threatening Grade 5: Death
Time Frame: During treatment (up to 5 years)
Measure: Number; unit: participants
Arm/Group | Arm I: Thal/ZLD | Arm II: ZLD
Number analyzed (Participants) | 35 | 33
participants | 17 | 13

ADVERSE EVENTS:
Arm/Group | Arm I: Thal/ZLD | Arm II: ZLD
Serious Adverse Events (participants affected / at risk) | 3/35 | 1/33
Other Adverse Events (participants affected / at risk) | 35/35 | 28/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Thal/ZLD (N=35) | Arm II: ZLD (N=33)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Infection without neutropenia (Infections and infestations) | 1 (2) | 0 (0)
Ureteral Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Thal/ZLD (N=35) | Arm II: ZLD (N=33)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (5)
Cardiovascular (Cardiac disorders) | 1 (1) | 0 (0)
Ischemia/Infarction (Cardiac disorders) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (3) | 0 (0)
Supraventricular arrhythmias (SVT/atrial fibrillation/flutter) (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Otitis External (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Vision (Eye disorders) | 0 (0) | 1 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 22 (189) | 6 (29)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 27 (133) | 20 (64)
Fever-No ANC (General disorders) | 1 (1) | 3 (3)
Pain (General disorders) | 2 (2) | 1 (1)
Rigors (General disorders) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infection without neutropenia (Infections and infestations) | 8 (12) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 1 (3) | 0 (0)
CPK (creatine phosphokinase) (Investigations) | 0 (0) | 1 (3)
Creatinine (Investigations) | 0 (0) | 2 (2)
Leukopenia (Investigations) | 3 (13) | 0 (0)
Lymphopenia (Investigations) | 2 (12) | 1 (1)
Neutropenia (Investigations) | 13 (59) | 2 (6)
Prothrombin Time (Investigations) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Ataxia (Nervous system disorders) | 2 (2) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 18 (48) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Ischemia-Cerebral (Nervous system disorders) | 1 (1) | 1 (1)
Neuro-Cranial (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 4 (5) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 28 (304) | 6 (10)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 3 (5) | 0 (0)
Tremor (Nervous system disorders) | 1 (3) | 1 (1)
Vasovagal Episode (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Ureteral Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 10 (24) | 8 (10)
Rash/dermatitis associated with high-dose chemotherapy or BMT studies. (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes